CLINICAL TRIAL: NCT01765387
Title: SPA THERAPY AS RECOVERY PROCEDURE AFTER EXERCISE: A PRAGMATIC CONTROLLED TRIAL
Brief Title: Spa Effects After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher in Physiotherapy, University of Malaga
Allocation: Non-Randomized | Model: Crossover | Masking: Single
Other Study IDs: FGEUGR01
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2013-01

CONDITIONS: Health Behavior
Keywords: Spatherpy; Aerobic exercise
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spa therapy (Experimental): A cycle of 3 Vichy shower and whirlpool baths are applied during 30-minutes period. Vichy sedative shower is applied for 90-120 sec to the sides of the trunk and the abdomen, avoiding as much as possible the gall bladder area, at a temperature of 36-38ºC. A short, partial jet spray followed the shower. A whirlpool bath is administered where subjects immersed the body until their clavicle level for a 10min period with a water temperature ranging 33.5-35.5 ºC. Aromatherapy application using lavender and chamomile oils is used in all Spa therapy sessions.
  Interventions: Behavioral: Spa session
- Control group (No Intervention): The control group perform a rest session in supine position in a room with neutral temperature condition with a same duration to Spa session. Participants of both groups are encouraged to drink water "ad libitum" to prevent dehydration.

INTERVENTIONS:
Behavioral: Spa session
  Arms: Spa therapy

SUMMARY:
The aim of this study is to evaluate the recovery effect of Spa therapy after aerobic exercise in cardiovascular, performance and perceived fatigue. A pragmatic controlled repeated measures, single-blind, trial is conducted. Thirty-four recreational sportspeople are required to visit a Sport-Centre and are assigned to a Spa-therapy or rest in a bed (control group) after complete a spinning session.

DETAILED DESCRIPTION:
Subjects perform the recovery session after completing the exercise protocol. Participants are allocated to the control or intervention group following an order of arrival to the study.

The spinning session is performed using the same protocol for all participants after 24h physical rest. They were asked to perform this session as a regular spinning class. The session is carried out in the afternoon (room temperature 22±3.5°C) on a modified spinning bike (Keiser®, M3). They are allowed to drink water during the session and performed the test, while they listen a compilation of music that lasted 50min composed of 9 tracks.

Each track corresponds to a specific phase of the spinning session. The phases being labeled as warm-up, sitting, seated climbing, jumping, and running, based on the official spinning program manual. Some phases are repeated during the session, the compilation being purposely designed for beginner practitioners of a spinning class. In addition to the music protocol, the participants are asked to maintain a pedal stroke cadence that had previously been established for each track. For the resistance applied to the flywheel, the participants are free to adjust it according to their sensation and interpretation of the spinning session.

Recovery Procedures

A cycle of 3 Vichy shower and whirlpool baths are applied during 30-minutes period. Vichy sedative shower are applied for 90-120 sec to the sides of the trunk and the abdomen, avoiding as much as possible the gall bladder area, at a temperature of 36-38ºC. A short, partial jet spray followed the shower. A whirlpool bath is administered where subjects immersed the body until their clavicle level for a 10min period with a water temperature ranging 33.5-35.5 ºC. Aromatherapy application using lavender and chamomile oils is used in all Spa therapy sessions.

The control group performed a rest session in supine position in a room with neutral temperature condition with a same duration to Spa session. Participants of both groups are encouraged to drink water "ad libitum" to prevent dehydration.

ELIGIBILITY:
Inclusion Criteria:

* 5-10 hours/wk of physical activity, no pharmaceutical drug intake in the past 3 months,
* No use of tobacco or other addictive substances,
* No pain symptoms from at least one year,
* No contradiction for high-intensity exercise following previous study about recovery after exercise

Exclusion Criteria:

* Signs or symptoms of medical disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
blood pressure | baseline, 5 minutes after spinning session, 5 minutes after recovery session

SECONDARY OUTCOMES:
heart rate | baseline, 5 minutes after spinning session, 5 minutes after recovery session
vertical jump test | baseline, 5 minutes after spinning session, 5 minutes after recovery session

OTHER OUTCOMES:
force handgrip | baseline, 5 minutes after spinning session, 5 minutes after recovery session
visual analogue scale fatigue | baseline,5 minutes after spinning session, 5 minutes after recovery session
body core temperature | baseline, 5 minutes after spinning session, 5 minutes after recovery session

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo Morales, PhD, Principal Investigator — University of Granada, Spain
Locations (1):
- Sport Club yo10, Granada, Granada, Spain

REFERENCES:
- [Derived] Cuesta-Vargas AI, Trave-Mesa A, Vera-Cabrera A, Cruz-Terron D, Castro-Sanchez AM, Fernandez-de-las-Penas C, Arroyo-Morales M. Hydrotherapy as a recovery strategy after exercise: a pragmatic controlled trial. BMC Complement Altern Med. 2013 Jul 18;13:180. doi: 10.1186/1472-6882-13-180. PMID 23866725